CLINICAL TRIAL: NCT00135603
Title: A Prospective Randomized Multicentric Trial Comparing Amoxicillin/Clavulanate Potassium Therapy to Appendectomy for Acute Non Complicated Appendicitis
Brief Title: Antibiotic Therapy Versus Appendectomy for Acute Appendicitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Corinne VONS, MD, PhD, Assistance Publique Hôpitaux de Paris
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P020915; AOR 02063
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-01

CONDITIONS: Appendicitis
Keywords: appendicitis.; adult.; treatment.; antibiotic therapy.; CT scanning.; randomized trial; safety
MeSH Terms: conditions — Appendicitis | interventions — Amoxicillin-Potassium Clavulanate Combination; Appendectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): appendectomy, actual usual treatment
  Interventions: Procedure: appendectomy
- B (Active Comparator): antibiotic therapy
  Interventions: Drug: amoxicillin/clavulanate potassium

INTERVENTIONS:
Drug: amoxicillin/clavulanate potassium — 1 gramme, 3 times a day, intra venous initially and then orally for one or two weeks
  Arms: B
Procedure: appendectomy — ablation of the appendix by laparotomy or laparoscopy
  Arms: A

SUMMARY:
The purpose of the study is to demonstrate that antibiotic therapy is as safe and effective as appendectomy for the treatment of acute non complicated appendicitis. Two hundred fifty patients will be included in a prospective multicentric randomized trial. The primary endpoint is the rate of intra abdominal infections in both therapeutic strategies. Other criteria will be studied including duration of hospital stay and absence from work during a follow up period of one year, parietal and abdominal complications and recurrent appendicitis after antibiotic therapy.

DETAILED DESCRIPTION:
Appendectomy is the most frequent intra-abdominal operation performed, accounting for the majority of admissions in a general surgery unit. Appendectomy has always been considered the cornerstone in the treatment of acute appendicitis.Nevertheless, the idea of a conservative treatment using antibiotics is not that recent. Current practices have proven the efficiency of antibiotic therapy in treating certain infectious abdominal conditions including: appendicular mass with or without periappendicular abscess and acute diverticulitis. This success has prompted the researchers to consider the exclusive use of antibiotic therapy in the treatment of non complicated appendicitis.

In patients with clinical suspicion of acute appendicitis (localized abdominal tenderness, inflammatory reaction...etc) a CT scan will be performed to confirm the diagnosis of non complicated appendicitis. This diagnosis is confirmed on the CT in the absence of any sign of either localized peritonitis, and/or perforation (extraluminal gas, appendicular abscess, or phlegmon).

After a thorough explanation of this study, the patient will be obliged to sign a written consent. Patients will be randomly assigned to either one of the two therapeutic modalities : an appendectomy,or an antibiotic treatment consisting of amoxicillin and clavulanate potassium.

This therapy will be continued until the normalisation of leucocytic count and C reactive protein are achieved. In order to demonstrate equivalent conclusive results comparing the two treatment modalities, the statistical consultant estimated the inclusion of at least 200 patients in the study. However, after considering the possible loss of a number of patients following their inclusion for a variety of reasons, it was decided that a total of 250 patients will be enrolled.

Rate of intra abdominal infections in both therapeutic strategies is the first endpoint to be compared. Duration of pain, diet, hospitalisation, absence from work will also be compared. In the group of patients treated by antibiotics, the rate of persistant and recurrent appendicitis after treatment will be evaluated. Recurrent appendicitis is not considered a complication as long as the recurrence of the appendicitis is uncomplicated. During the followup period of one year, long-term complications will be observed including: abdominal hernia, adhesive intestinal occlusion, and others.

ELIGIBILITY:
Before CT scanning

Inclusion Criteria:

* Clinical suspicion of appendicitis
* Age more than 18 years

Exclusion Criteria:

* Clinical signs of generalized peritonitis
* Previous take of antibiotics within the 5 days preceding the presentation
* Allergy or intolerance to lactamases and/or clavulanate potassium
* Corticosteroid or anticoagulant therapy
* Patient with a known inflammatory bowel disease (Crohn's disease or ulcerative colitis)
* Pregnant women
* Patient with iode allergy
* Renal insufficiency (creatinine > 200 )

CT scanning:

Inclusion Criteria:

* Appendix diameter > 6 mm

Exclusion Criteria:

* Appendix non visualised
* Signs of localized peritonitis:

  * extradigestive gas
  * fluid collection around the appendix
  * generalized intraperitoneal fluid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2004-02; Primary Completion 2008-02 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
rate of intra abdominal infections in both therapeutic strategies | 30 days

SECONDARY OUTCOMES:
duration of pain | 30 days
duration of hospitalisation | 30 days
duration of absence from work | 30 days
rate of wound infection | 30 days
recurrence of appendicitis | 12 months
rate of abdominal hernia | 12 months
rate of adhesive intestinal occlusion | 12 months
cost | 30 days and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Vons, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (5):
- France (5):
  - Antoine Béclère Hospital - Department of Surgery, Clamart
  - Henri Mondor Hospital, Créteil
  - Hotel Dieu Hospital, Department of Digestive Surgery, Paris
  - Cochin Hospital, Department of Digestive Surgery, Paris
  - Lariboisière Hospital, Department of Digestive Surgery, Paris

REFERENCES:
- [Derived] Vons C, Barry C, Maitre S, Pautrat K, Leconte M, Costaglioli B, Karoui M, Alves A, Dousset B, Valleur P, Falissard B, Franco D. Amoxicillin plus clavulanic acid versus appendicectomy for treatment of acute uncomplicated appendicitis: an open-label, non-inferiority, randomised controlled trial. Lancet. 2011 May 7;377(9777):1573-9. doi: 10.1016/S0140-6736(11)60410-8. PMID 21550483